CLINICAL TRIAL: NCT06394726
Title: Investigation of the Effects of Aerobic and Core Stabilization Exercises on Primary Dysmenorrhea in High School Female Students
Brief Title: Examining the Impact of Aerobic and Core Exercises on Primary Dysmenorrhea in High School Females
Acronym: Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, AYCAN ÇAKMAK REYHAN, Principal Investigator, Istanbul Bilgi University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: İstanbulBilgiiiU
Record Dates: First submitted 2024-02-26; First posted 2024-05-01 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Dysmenorrhea
Keywords: Aerobic exercise; Core Stabilization Exercises
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (Active Comparator): Aerobic Exercise Group For 3 months, participants will engage in a total of 150 minutes of exercise per week, either 30 minutes for 5 days a week or 50 minutes for 3 days a week.
  Interventions: Behavioral: Exercise İntervention
- Core Stabilization Exercise Group (Active Comparator): Core Stabilization Exercise Group for 3 months, 2 sets of exercises, each comprising 10 repetitions per set.
  Interventions: Behavioral: Exercise İntervention

INTERVENTIONS:
Behavioral: Exercise İntervention — Aerobic and Core Stabilization Exercise Intervention

SUMMARY:
Dysmenorrhea, derived from ancient Greek, translates to 'difficult monthly flow' and refers to painful cramps during menstruation, a common cause of pelvic pain. The pain, often in the lower abdomen, results from uterine pressure exceeding 60 mmHg. Symptoms include suprapubic pain, radiating discomfort, nausea, diarrhea, and headache, impacting quality of life. Etiology involves factors like age at menarche, heavy flow, lifestyle, and medical conditions.

Dysmenorrhea is categorized as primary (without underlying pathology) or secondary (due to conditions like endometriosis). Its prevalence is high in adolescence, affecting daily life, school, and health. Research aims to assess how aerobic and core exercises influence pain and quality of life in adolescent females (14-18 years). Participants are randomly assigned to study and control groups, exploring the potential benefits for health, well-being, and academic performance.

DETAILED DESCRIPTION:
Dysmenorrhea, which begins approximately 1-2 years after the start of menstruation in women, continues until the 40s, although it shows its effects more in adolescent female students between the ages of 18-25. Dysmenorrhea pain, which is seen intermittently in the form of contractions and cramps, is usually in the middle of the highest intensity value. It is also emphasized that dysmenorrhea has important economic consequences. It has been reported that the total healthcare costs of patients with primary dysmenorrhea are greater than the healthcare costs of women without dysmenorrhea. In Japan, the total healthcare costs of patients with primary dysmenorrhea were reported to be 2.2 times greater than the healthcare costs of women without dysmenorrhea after adjusting for baseline characteristics. Although dysmenorrhea is not a life-threatening condition, it can cause a significant burden on individuals and communities, greatly affecting quality of life and well-being. Both aerobic and core exercises reduce the severity of dysmenorrhea, especially at young ages. It has been proven that core exercises are an effective non-pharmacological method to reduce pain and are a cost-free pain-reducing practice. Aerobic exercises are exercises that increase cardiopulmonary endurance capacity by activating the circulatory and respiratory systems through rhythmic and dynamic contraction of large muscle groups. In this study, a brisk walking program, which is a type of aerobic exercise, will be created for adolescent students and its effects on primary dysmenorrhea will be evaluated. Studies on this subject have concluded that aerobic exercise has an effect on some menstrual symptoms of adolescent high school female students, and that dysmenorrhea and heavy menstrual bleeding can be controlled or prevented by performing these exercises regularly and continuously. Secondly, it has also been found that aerobic exercises are positively related to the information processing efficiency, attention, memory and cognitive control of adolescents. Although there is limited evidence, it is thought that physical activity can have a positive effect on improving academic performance, cognitive abilities and mental functions in children. It has also been reported that aerobic exercises have a protective effect against the risk of diseases (childhood obesity, asthma, etc.) by keeping the heart rate and weight control low and improving cardiovascular health. Regular aerobic exercises, especially in adolescents; It leads to hormonal changes by increasing functional work capacity, daily life activity level and quality of life in individuals with systematic diseases and reducing psychological stress. These hormonal changes include the fact that aerobic exercises increase the release of endorphins. Increased endorphin release causes an increase in pain threshold. For this reason, by reducing dysmenorrhea pain with the aerobic and core exercises will use in the study; It is aimed to increase the quality of life of high school-aged adolescents by increasing the duration of class attendance, drug-free pain control, desire to study, socialization and exam success, and to improve adolescent health with applications in the field of physiotherapy. The core can be defined as the trunk or the region that provides the connection between the legs and arms. This region, which is mentioned as the central region of the body, is the point where the stabilization of the abdominal, paraspinal and gluteal muscles, consisting of the muscles, nerves, skeleton and other connective tissues that form the spine, pelvis, abdominal cavity and upper structures, is critical for optimal performance and is also defined as the lumbopelvic region. Core exercises are; These are exercises that include exercises to train the muscles that control and stabilize the movements of the abdominal, lumbar and gluteal regions. Core exercises are exercises that help increase muscle balance and strength. These exercises play an active role in ensuring that muscles move correctly. Strengthening the core area is important not only for sports performance but also for maintaining proper body posture. These exercises aim to control balance, improve upper extremity functions, ensure proper posture, increase stabilization, and minimize pain in the pelvic and abdominal areas. The reason why investigators chose this topic is that although there are studies in the literature evaluating the effects of core and aerobic exercises separately on dysmenorrhea, there are no studies on the effects of these two exercises on dysmenorrhea with a combined program. In addition, as the negative effects of menstrual pain on high school-age young people are seen as a normal problem, this causes an increase in the number of primary dysmenorrhea cases, an increase in the use of pharmacological supplements, and a negative impact on the psychological and social quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Be nulliparous (have not given birth) and be between the ages of 14-18.
* Volunteer to participate.
* Have no active sexual life.
* Have a regular menstrual cycle.
* Report a pain intensity of 5 or above on the Visual Analog Scale (VAS).
* Have a Body Mass Index (BMI) between 19 and 24.9.
* Not have polycystic ovary syndrome or undergone any surgical operation related to female diseases.
* Not engage in regular exercise.
* Not have any chronic, systemic, neurological, or endocrinological diseases.

Exclusion Criteria:

* Participate in tele-rehabilitation and exercise diary for less than 3 days.
* Use an intrauterine device.
* Have taken pharmacological supplements in the last 3 months or during the study tracking period (due to reasons such as flu, COVID, etc.).
* Have any physical impediment restricting physical activity.

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 50 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | baseline and 12 weeks
  VAS is a common tool for assessing subjective experiences like pain or mood intensity. It consists of a 10-centimeter line with clear endpoints representing extreme sensations. Participants mark a point on the line corresponding to their perception, such as "No Pain" to "Worst Pain Imaginable." The distance from "No Pain" provides a quantitative measure. Easy to administer and adaptable, VAS is widely used in clinical and research settings for various subjective states beyond pain, requiring no specialized training. "In this scale, '0' corresponds to the best, and '10' to the worst
Functional and Emotional functional and emotional measure of dysmenorrhea (FEMD) | baseline and 12 weeks
  "FEMD" stands for Functional and Emotional Measure of Dysmenorrhea. Dysmenorrhea refers to painful menstruation, commonly known as menstrual cramps. The FEMD is a tool or scale used to assess both the functional and emotional impacts of dysmenorrhea on individuals. The functional aspect of the FEMD typically evaluates the severity of physical symptoms associated with dysmenorrhea, such as the intensity of pain, its duration, any associated symptoms like nausea or vomiting, and how these symptoms affect daily activities or functioning. The scale consists of 14 items and 2 subscales. Each item is scored on a scale from 1 to 5: (1) Not at all like my condition, (2) Not much like my condition, (3) Somewhat like and somewhat unlike my condition, (4) Much like my condition, (5) Very much like my condition. There are no reverse items. As scores increase on this scale, individuals' levels of functional and emotional impact from dysmenorrhea also increase."

SECONDARY OUTCOMES:
SF-36 Short Form 36 Health Survey | baseline and 12 weeks
  The S-F36 Health Survey is a widely used questionnaire for assessing health-related quality of life. It measures 8 health concepts: physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations, and mental health. These concepts are grouped into two dimensions: physical health and mental health. Scoring is based on responses to each question in each subscale, typically ranging from 0 to 100. Higher scores indicate better perceived physical functioning
A dysmenorrhea monitoring form | baseline and 12 weeks
  A dysmenorrhea monitoring form typically includes various aspects related to menstrual pain and associated symptoms. Here's an example of a dysmenorrhea monitoring form.
Dysmenorrhea Impact Scale short form | baseline and 12 weeks
  The "Dismenorrhea Impact Scale" is a tool used to assess the functional and emotional symptoms associated with dysmenorrhea (menstrual pain). This scale evaluates individuals' limitations in daily life activities and the emotional distress they experience due to menstrual pain.This scale serves as an important tool in determining the impact of menstrual pain on individuals' quality of life and in developing appropriate treatment strategies.The scale does not contain reverse items. It is a five-point Likert scale, scored as follows: Strongly Disagree (1), Disagree (2), Neutral (3), Agree (4), Strongly Agree (5). The first 8 items belong to the cognitive/emotional subscale, while the last 5 items fall within the physiological subscale.
Menstrual Symptom Questionnaire | baseline and 12 weeks
  MAS is a tool used to assess individuals' attitudes towards menstruation. It measures beliefs, feelings, and behaviors related to menstruation. The scale typically consists of a series of statements or items, to which individuals respond based on their agreement or disagreement.Due to the difficulty in adapting the original 7-point Likert scale assessment form into Turkish, the Turkish version of the scale has been converted to a 5-point evaluation form ranging from 1 to 5 (1. Strongly Disagree, 2. Disagree, 3. Neutral, 4. Agree, 5. Strongly Agree). Higher average scores obtained from items, subgroups, or the entire scale indicate a "positive" attitude towards menstruation.

CONTACTS AND LOCATIONS:
Overall Officials: Aycan Cakmak Reyhan, PhD, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No